CLINICAL TRIAL: NCT03691857
Title: Evaluation of the Feasibility and Accuracy of an Ultrasound Algorithm for Acute Dyspnea Diagnosis in the Emergency Department
Brief Title: Feasibility and Accuracy of an Ultrasound Algorithm for Acute Dyspnea Diagnosis in the Emergency Department
Acronym: EMERALD-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHOUIHED Tahar (Other)
Responsible Party: Sponsor-Investigator, CHOUIHED Tahar, Study chair, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A02136-49
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute non-traumatic dyspnea patients (Other): Patients with acute non-traumatic dyspnea managed in the emergency department to assess the diagnostic accuracy of an ultrasound algorithm (EMERALD-US) dedicated to emergencies using lung, cardiac and vascular ultrasound for the 3 main dyspnea causes (heart failure, pneumonia and obstructive pulmonary disease exacerbation)
  Interventions: Procedure: Ultrasound algorithm (EMERALD-US)

INTERVENTIONS:
Procedure: Ultrasound algorithm (EMERALD-US) — Ultrasound algorithm EMERALD-US is an dedicated to emergencies using lung, cardiac and vascular ultrasound for the 3 main dyspnea causes (heart failure, pneumonia and obstructive pulmonary disease exacerbation) in patients with acute non-traumatic dyspnea managed in the emergency department. The ultrasounds will be performed within first hour after first medical contact in emergency department by another emergency physician not in charge of the patient. The ultrasound results will be not shared with the emergency physician in charge of the patient.

SUMMARY:
The management of chest pain has revolutionized its prognosis, primarily by improving urgent diagnosis of myocardial infarction. Currently, acute dyspnea is twice as frequent as chest pain and its associated mortality is much higher (16% of acute dyspnea admitted to emergency departments (ED) ).

Inappropriate treatment of acute dyspnea in the ED is frequent (30%) and is associated with a tripling of intra-hospital mortality after adjustment for confounding factors (2.83, IC 1.48 to 5.41, p=0.002). Other elements have also highlighted the importance of a quick and appropriate acute dyspnea diagnosis:

* The 2015 European Guidelines on acute heart failure emphasize the need for appropriate treatment within 90 minutes after the first medical contact.
* Inadequate treatment of chronic bronchitis decompensation is associated with a doubling of intra-hospital mortality.
* An initiation of antibiotic treatment within 4 hours of admission for pneumonia is recommended.
* 30% of pulmonary embolisms are not diagnosed during the initial emergency department visit, whereas their mortality in the absence of treatment is 25%.

Lung, venous and (simplified) cardiac ultrasound is associated with improved diagnostic performance in ED. However, no ultrasound algorithm dedicated to emergency physicians has been formally validated. The Blue Protocol (Lichtenstein et al., Chest 2008) has been validated in intensive care patients with very different phenotypes than those admitted to the ED. Pivetta et al. (Chest 2015) proposed an algorithm focused solely for the diagnosis of heart failure, thus not providing a diagnosis for all the other causes of dyspnea in ED. Finally, Zanbonetti et al. (Chest 2017) proposed an "unguided" ultrasound use, notably integrating inferior vena cava evaluation. However, measuring the inferior vena cava is difficult at the start of ED management when patients are in acute respiratory distress.

DETAILED DESCRIPTION:
The investigators aim to assess the feasibility and accuracy of a new pragmatic and original ultrasound algorithm adapted for acute dyspnea diagnosis in the emergency department.

This primary objective of this prospective multicenter study is to assess the diagnostic accuracy of an ultrasound algorithm (EMERALD-US) dedicated to emergencies using lung, cardiac and vascular ultrasound for the 3 main dyspnea causes (heart failure, pneumonia and obstructive pulmonary disease exacerbation) in patients with acute non-traumatic dyspnea managed in the emergency department. Ultrasound exams will be blindly read by a centralized core laboratory after the standardized acquisition of all exams by a physician not involved in the care of patients in the ED. The main discharge diagnosis from initial hospitalization (heart failure, pneumonia and obstructive pulmonary disease exacerbation) will be adjudicated by a college of 3 senior physicians (emergency physician, cardiologist and internist) blinded to the use of ultrasound in the ED.

The secondary objectives of the study are to:

A/ Assess the feasibility of the ultrasound algorithm (EMERALD-US) in emergency departments.

B/ Assess the association between the diagnosis obtained from the ultrasound algorithm (EMERALD-US) and the results of additional (laboratory and radiological exams.

C/ Assess the diagnostic accuracy of the ultrasound algorithm (EMERALD-US) for less frequent dyspnea causes (pulmonary embolism, pleural effusion).

D/ Assess, the diagnostic accuracy of clinical (including BREST and PREDICA score), laboratory and radiological variables.

E/ Assess, the improvement in diagnosis accuracy with the ultrasound algorithm (EMERALD-US) on top of the diagnostic accuracy of clinical, laboratory and radiological exams.

F/ Assess the association between misdiagnosis (without using ultrasound) and survival at D30.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years old
* Patients with non-traumatic acute dyspnea managed in the emergency department
* Patients affiliated with a social security system

Exclusion Criteria:

* Patients in cardiac arrest
* Patients in persistent shock
* Patients with impaired consciousness (Glasgow Score<9)
* Patients with a history of thoracic surgery or pulmonary fibrosis
* Dementia
* Patients with Acute Coronary Syndrome with ST elevation
* Known current pregnancy
* Patients under guardianship, trusteeship or legal protection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Main discharge diagnosis (heart failure, pneumonia and obstructive pulmonary disease exacerbation) | an average of 2 weeks (from date of admission in the emergency department until the date of hospitalization discharge)
  Main discharge diagnosis (heart failure, pneumonia and obstructive pulmonary disease exacerbation) adjudicated by a college of 3 senior physicians (emergency physician, cardiologist and internist) blinded to the use of ultrasound in the emergency department

SECONDARY OUTCOMES:
Duration of the ultrasound examination | up to 30 minutes
  Duration of the ultrasound examination is defined by the delay between the first and last contact between the ultrasound probe and the patient
Proportion of complete realization of the ultrasound algorithm | up to 30 minutes
  Proportion of complete realization of the ultrasound algorithm through study completion
Diagnosis given by the algorithm after core-lab reading of the blinded ultrasound compared to the diagnosis provided by the emergency physician based on the EMERALD algorithm in the emergency department | At baseline
  Diagnosis given by the algorithm after core-lab reading of the blinded ultrasound compared to the diagnosis provided by the emergency physician based on the EMERALD algorithm in the emergency department
Patient management time in the emergency department | An average of 24 hours (Time between the time of entry to the emergency department and the time of discharge).
  Patient management time in the emergency department is defined by the time between the time of entry to the emergency department and the time of discharge specified in the patient's medical report.
Brain Natriuretic Peptide (BNP) or N-terminal pro-brain natriuretic peptide concentration | At admission in the emergency department
  Assess the association between the diagnosis obtained from the ultrasound algorithm (EMERALD-US) and the results of additional laboratory exams. NT pro BNP will be measured from the biobanking.
C Reactive protein and procalcitonin concentration, | At admission in the emergency department
  Assess the association between the diagnosis obtained from the ultrasound algorithm (EMERALD-US) and the results of additional local laboratory exams
D-dimer concentration, | At admission in the emergency department
  Assess the association between the diagnosis obtained from the ultrasound algorithm (EMERALD-US) and the results of additional local laboratory exams
Radiological diagnosis (chest X-ray or chest CT). | At admission in the emergency department
  Assess the association between the diagnosis obtained from the ultrasound algorithm (EMERALD-US) and the results of additional local radiological exams
Main discharge diagnosis including combined diagnosis (e.g. heart failure and pneumonia) from initial hospitalization adjudicated by a college of 3 senior physicians | An average of 2 weeks (from date of admission in the emergency department until the date of discharge)
  Main discharge diagnosis including combined diagnosis (e.g. heart failure and pneumonia) from initial hospitalization adjudicated by a college of 3 senior physicians
All-cause mortality at D30. | At Day 30
  Assess the association between misdiagnosis (without using ultrasound) and survival at D30

CONTACTS AND LOCATIONS:
Overall Officials: Tahar CHOUIHED, MD, Principal Investigator — Central Hospital, CHRU de Nancy, France; Nicolas GIRERD, MD PhD, Study Chair — CHRU de Nancy, France; Patrick ROSSIGNOL, MD PhD, Study Chair — CHRU de Nancy, France
Locations (7):
- France (7):
  - CH de Chalons en Champagne, Châlons-en-Champagne
  - Hôpital Simone Veil, Eaubonne
  - CHRU Nancy, Nancy
  - AP-HP - Hôpital Cochin, Paris
  - AP-HP - Hôpital Lariboisière, Paris
  - CH de Sarreguemines, Sarreguemines
  - CHRU de Strasbourg, Hôpital de Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaeger D, Duchanois C, Duarte K, Lepage X, Merckle L, Bassand A, Buessler A, Chauvin A, Bokobza J, Penine A, Giacomin G, Brossard C, Girerd N, Chouihed T. Performance of an ultrasound diagnostic algorithm for acute dyspneic patients in the emergency department: an EMERALD-US protocol. BMJ Open. 2025 Aug 10;15(8):e101432. doi: 10.1136/bmjopen-2025-101432. PMID 40784781